CLINICAL TRIAL: NCT07262502
Title: EVALUATION OF THE CLINICAL SUCCESS OF A HYDROPHILIC FISSURE SEALANT APPLIED TO LOWER PERMANENT MOLARS UNDER DRY AND WET CONDITIONS
Brief Title: Evaluation of the Clinical Success of Hydrophilic Fissure Sealants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Mehmet Ünal, PhD, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24.DUS.010
Record Dates: First submitted 2025-11-23; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pit and Fissure Caries (Disorder); Pit and Fissure Sealants
Keywords: pit and fissure sealants; Preventive Dentistry
MeSH Terms: conditions — Van der Woude syndrome | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pit and fissure sealant treatment (Experimental)
  Interventions: Other: pit and fissure sealant

INTERVENTIONS:
Other: pit and fissure sealant — For each tooth to be treated with pit and fissure sealant, phosphoric acid will be used for pre-treatment. One group will be dried with an air-water spray for 3 seconds, while the drying time for the other group of teeth in the opposing jaw will be 15 seconds.

SUMMARY:
The study group will consist of children aged 7-11 years who are systemically healthy and who apply to the Pediatric Dentistry Clinic of the Faculty of Dentistry, Afyonkarahisar Health Sciences University for routine dental treatment.

In the study, fissure sealants will be applied to the first molars with opposing deep pits and fissures in the same jaw.

The study will involve the application of fissure sealants to the first molars with opposing deep pits and fissures in the same jaw.

It was decided to include a total of 500 teeth from 250 patients in the study, with 250 teeth in each group.

The occlusal surface of each tooth will be dried and etched with 37% phosphoric acid (Eco-Etch; Ivoclar Vivadent, Inc. Schaan, Liechtenstein) and thoroughly rinsed for 30 seconds.

If saliva contamination occurs, the surface will be etched again. The treated tooth will be air-dried for 3 seconds and the tooth in the opposing jaw for 15 seconds. Subsequently, the relevant fissure sealant (Pulpdent, Embrace Wetbond Pit and Fissure Sealant) will be applied to the occlusal surface of each tooth and cured for 20 seconds using a light-curing unit at an intensity of 500 mW/cm².

After restoration, articulation paper will be used to check for any high spots in the occlusion; if found, excess material will be removed using a finishing bur.

Clinical evaluations of marginal integrity, marginal color change, and retention after the liner is placed will be performed at 3, 6, 9, and 12 months using the World Health Organization probe according to the Ryge and Synder criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 7-11 who applied for dental examination at the Department of Pediatric Dentistry, Faculty of Dentistry, Afyon Health Sciences University.

  2. Patients must be systemically healthy and have no mental or physical disabilities.

  3. Permanent first molars must be fully erupted in the mouth, and at least 3 first molars must be indicated for non-invasive fissure sealant application (having narrow, deep fissures prone to decay).

  4. Permanent first molars to receive fissure sealants must not have hypomineralized areas such as fluorosis or first molar incisal hypomineralization.

  5. Permanent first molars must not have occlusal or approximal caries.

Exclusion Criteria:

* 1. Patients must not be between the ages of 7 and 11. 2. Patients must not be systemically healthy and must have no mental or physical disabilities.

  3. Patients must have poor oral hygiene. 4. There must be caries in the permanent first molars where fissure sealants will be applied.

  5. Presence of hypomineralized areas such as fluorosis or first molar hypomineralization on the permanent first molars where fissure sealants will be applied.

  6. Patients not cooperating with the procedures to be performed. 7. Patients or their parents not wanting to participate in the study.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Edge discoloration | 3-6-9-12 months
  A: No color change between the restoration and the tooth structure B: Localized, mostly removable superficial color change C: Pulpal discoloration

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided